CLINICAL TRIAL: NCT01726335
Title: An Open-Label Study of Oral Antipsychotics Replacement by Prolonged Release Risperidone (Risperdal Consta) in Schizophrenic Subjects With Bad Adhesion to the Treatment
Brief Title: Switching From Oral Antipsychotics to Long-Acting Risperidone in Participants With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012484; RISSCH4135
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Results first posted 2013-07-24 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Risperdal consta
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Risperidone prolonged release (Experimental): Risperidone will be administered as intramuscular injection as 25 milligram (mg) every two weeks, from Week 1 to 50, wherein after Week 3, dose may be adjusted up to 50 mg at physician criterion. For first two weeks, previous oral antipsychotic drug will be maintained and the dose will be gradually decreased and will cease at Week 3.
  Interventions: Drug: Risperidone prolonged release

INTERVENTIONS:
Drug: Risperidone prolonged release — Risperidone will be administered as intramuscular injection as 25 milligram (mg) every two weeks, from Week 1 to 50, wherein after Week 3, dose may be adjusted up to 50 mg at physician criterion. For first two weeks, previous oral antipsychotic drug will be maintained and the dose will be gradually decreased and will cease at Week 3.
  Other Names: - Risperdal consta

SUMMARY:
The purpose of this study is to evaluate efficacy, safety and tolerance of long-acting risperidone when switching from oral antipsychotics in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-centric (conducted in more than one center) and non-comparative study of long-acting risperidone in participants with schizophrenia who have a previous history (in the last 12 months) of bad adherence to the oral antipsychotic treatment of first or second generation. The duration of this study will be 24 weeks and will include following visits: Screening, Baseline, Week 2, 4, 8, 12, 16, 20, 24, 38 and 50 (End visit or early withdrawal). All the eligible participants (after risperidone intolerance test during screening) will receive a dose of 25 milligram risperidone every two weeks by intramuscular injection (injection of a substance into a muscle). Efficacy and safety of the participants will primarily be evaluated by Positive and Negative Syndromes Scale and Extrapyramidal Symptom Rating Scale, respectively. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have schizophrenia diagnosis by Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV)
* Be on treatment with oral antipsychotic of first or second generation, for a minimum time of 12 months
* Previous history of bad adhesion to oral antipsychotic treatment in the last 12 months
* Total Positive and Negative Syndrome Scale score less than or equal to 90, the conceptual disorganization, hallucinatory behavior, suspicion and not usual content of thought must be less than or equal to 4
* Be not pregnant as showed on negative pregnancy serum test

Exclusion Criteria:

* Contraindication or known hypersensitivity to risperidone
* Previous history of unsatisfactory response to risperidone
* Previous history of refractivity to the other second generation antipsychotics
* Use of antipsychotic of intramuscular deposit in the last 12 months
* Other mental disturbances of DSM-IV axis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical trial, Study Director — Janssen-Cilag Ltd.
Locations (5):
- Brazil (5):
  - Curitiba
  - Porto Alegre
  - Rio de Janeiro
  - Salvador
  - São Paulo

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone Prolonged Release: Risperidone was administered as an intramuscular injection (injection of a substance into a muscle) at a dose of 25 milligram (mg), every two weeks, from Week 1 to 50, wherein after Week 3, dose was adjusted up to 50 mg at Physician criterion. For first two weeks, previous oral antipsychotic drug was maintained and the dose was gradually decreased and ceased at Week 3.
Period: Overall Study
Arm/Group | Risperidone Prolonged Release
Started | 53
Completed | 29
Not Completed | 24
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 15
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 2
Not completed — Exacerbation of psychotic symptoms | 1

BASELINE CHARACTERISTICS:
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 39
Positive and Negative Syndromes Scale (PANSS) Total Score [Mean (Standard Deviation); unit: Units on a scale] — The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
  Units on a scale | 58.80 (1.82)

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndromes Scale (PANSS) Total Score at Week 2
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
Time Frame: Week 2
Population: Intent-to-treat-efficacy evaluation (ITTe) population included all the Participants who received at least one dose of study medication and provided one measure post-baseline of efficacy.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 51
Units on a scale | 55.53 (1.82)

2. Primary Outcome: Positive and Negative Syndromes Scale (PANSS) Total Score at Week 4
Description: as for outcome 1
Time Frame: Week 4
Population: The ITTe population included all the Participants who received at least one dose of study medication and provided one measure post-baseline of efficacy.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 51
Units on a scale | 53.82 (1.83)

3. Primary Outcome: Positive and Negative Syndromes Scale (PANSS) Total Score at Week 8
Description: as for outcome 1
Time Frame: Week 8
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 51
Units on a scale | 51.28 (1.86)

4. Primary Outcome: Positive and Negative Syndromes Scale (PANSS) Total Score at Week 16
Description: as for outcome 1
Time Frame: Week 16
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 51
Units on a scale | 50.55 (1.98)

5. Primary Outcome: Positive and Negative Syndromes Scale (PANSS) Total Score at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 51
Units on a scale | 48.95 (2.13)

6. Secondary Outcome: Clinical Global Impressions (CGI) - Disease Severity Score
Description: The CGI rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 indicates to "normal, not at all ill" and a rating of 7 indicates "among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Baseline and Week 2, 4, 8, 16, 24, 38 and 50
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 51
Units on a scale
  Baseline | 3.55 (0.13)
  Week 2 | 3.37 (0.13)
  Week 4 | 3.30 (0.13)
  Week 8 | 3.21 (0.13)
  Week 16 | 3.10 (0.14)
  Week 24 | 2.92 (0.15)
  Week 38 | 2.94 (0.15)
  Week 50 | 3.19 (0.16)

7. Secondary Outcome: Extrapyramidal Symptoms Rating Scale (ESRS) Total Score
Description: The ESRS is used to assess four types of drug-induced movement disorders administered as a questionnaire. Score range from 0 to 6 (0 is absent and 6 is extremely severe).
Time Frame: Baseline and Week 2, 4, 8, 16, 24 and 50
Population: Intent-to-treat-safety evaluation (ITTs) population included all the Participants who received at least one dose of study medication and were reassessed after the start of use. 'N' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 50
Units on a scale
  Baseline | 0.460 (0.073)
  Week 2 | 0.416 (0.072)
  Week 4 | 0.272 (0.073)
  Week 8 | 0.289 (0.074)
  Week 16 | 0.271 (0.079)
  Week 24 | 0.221 (0.082)
  Week 50 | 0.089 (0.086)

8. Secondary Outcome: Drug Attitude Inventory (DAI-10)
Description: The DAI-10 is a 10-item questionnaire to assess 1) subjective experience of drug and 2) attitudes and beliefs toward neuroleptics which may influence compliance in schizophrenia participants. It is the binary scale assessing the participant's subjective response. A 'compliant' response is scored as +1; a dysphoric response is scored as -1. A positive sum of items indicates a positive subjective response (SR); a negative sum of scores indicates a negative SR (non-compliant). The final score is the grand total of the positive and negative points. Total score ranges from (-) 10 to (+) 10, higher score indicates positive SR (compliant) and lower score indicates negative SR (non-compliant).
Time Frame: Screening, and Week 8, 24 and 50
Population: ITTs population included all the Participants who received at least one dose of study medication and were reassessed after the start of use. 'N' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 51
Units on a scale
  Screening | 2.78 (0.62)
  Week 8 | 4.45 (0.64)
  Week 24 | 4.59 (0.69)
  Week 50 | 5.07 (0.77)

9. Secondary Outcome: Short Form-36 (SF-36) - Quality of Life
Description: The SF-36 is a survey of participant health. It consists of eight scaled scores, which are the weighted sums of the questions in their section. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Each item is scored on a 0-100 range so that the lowest and highest possible scores are set at 0 and 100, respectively. All items are scored so that a high score defines a more favorable health state.
Time Frame: Baseline and Week 50
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 51
Units on a scale
  Functional capacity : Baseline | 79.2 (21.4)
  Physical aspect : Baseline | 48.2 (40.2)
  Pain : Baseline | 73.7 (27.2)
  Health General State : Baseline | 60.7 (18.4)
  Vitality : Baseline | 53.8 (21.2)
  Social Aspect : Baseline | 56.1 (28.0)
  Emotional Aspect : Baseline | 34.9 (38.4)
  Mental Health : Baseline | 58.9 (21.9)
  Functional capacity : Week 50 | 67.9 (31.6)
  Physical aspect : Week 50 | 52.9 (41.3)
  Pain : Week 50 | 75.4 (29.5)
  Health General State : Week 50 | 62.7 (19.5)
  Vitality : Week 50 | 53.1 (18.3)
  Social Aspect : Week 50 | 59.9 (26.2)
  Emotional Aspect : Week 50 | 55.0 (41.7)
  Mental Health : Week 50 | 56.6 (20.6)

10. Primary Outcome: Positive and Negative Syndromes Scale (PANSS) Total Score at Week 38
Description: as for outcome 1
Time Frame: Week 38
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 51
Units on a scale | 47.40 (2.26)

11. Primary Outcome: Positive and Negative Syndromes Scale (PANSS) Total Score at Week 50
Description: as for outcome 1
Time Frame: Week 50
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 51
Units on a scale | 49.72 (2.32)

12. Secondary Outcome: Personal and Social Performance (PSP) Scale Score
Description: The PSP scale assesses the degree of a participant's dysfunction (ranging from i [absent] to vi [very severe) within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, disturbing and aggressive behavior. The overall score ranges from 1 to 100. Based on the 4-domains there was one total score. Participants with a score of 71 to 100 had a mild degree of difficulty; from 31 to 70, varying degrees of disability; participants with scores of 30 or less function so poorly as to require intensive supervision.
Time Frame: Screening, and Week 8, 16, 24, 38 and 50
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 34
Units on a scale
  Screening | 60.0 (2.9)
  Week 8 | 66.4 (2.4)
  Week 16 | 72.6 (2.3)
  Week 24 | 71.7 (2.1)
  Week 38 | 71.8 (2.1)
  Week 50 | 69.1 (2.2)

13. Secondary Outcome: Global Assessment of Functioning (GAF) Scale Score
Description: The GAF scale is a 100-point tool rating overall psychological, social and occupational functioning of adults. The higher score range (91-100) refers to a superior functioning in a wide range of activities, and absence of symptoms. The lower score range (1-10) refers to persistent danger of severely hurting self or others; or persistent inability to maintain minimum personal hygiene; or serious suicidal act with clear expectation of death.
Time Frame: Screening, and Week 8, 16, 24, 38 and 50
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Risperidone Prolonged Release
Number analyzed (Participants) | 34
Units on a scale
  Screening | 62.6 (3.1)
  Week 8 | 67.5 (2.6)
  Week 16 | 72.5 (2.5)
  Week 24 | 71.4 (2.3)
  Week 38 | 73.9 (2.3)
  Week 50 | 68.6 (2.3)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 50
Description: Intent-to-treat-safety evaluation (ITTs) population included all the Participants who received at least one dose of study medication and were reassessed after the start of use.
Arm/Group | Risperidone Prolonged Release
Serious Adverse Events (participants affected / at risk) | 3/53
Other Adverse Events (participants affected / at risk) | 40/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone Prolonged Release (N=53)
Psychomotor hyperactivity (Nervous system disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone Prolonged Release (N=53)
Hyperprolactinaemia (Endocrine disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Salivary hypersecretion (Gastrointestinal disorders) | 1
Application site pain (General disorders) | 1
Asthenia (General disorders) | 1
Feeling jittery (General disorders) | 1
Irritability (General disorders) | 2
Oedema (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Influenza (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood prolactin increased (Investigations) | 6
Blood thyroid stimulating hormone increased (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Akathisia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dystonia (Nervous system disorders) | 2
Extrapyramidal disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Sedation (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 4
Apathy (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Fear (Psychiatric disorders) | 1
Hostility (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 12
Orgasm abnormal (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 3
Schizophrenia, disorganised type (Psychiatric disorders) | 4
Amenorrhoea (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 2
Erectile dysfunction (Reproductive system and breast disorders) | 1
Galactorrhoea (Reproductive system and breast disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the Principal Investigator is that the Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the Sponsor for review. The Sponsor can require changes to the communication and can extend the embargo.